CLINICAL TRIAL: NCT01842087
Title: An Investigation Into Pulse Fiber Fermentation and Nitrogen Excretion in Patients With Chronic Renal Failure
Brief Title: The Effects of Fiber Fortified Foods to the Diets of Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Saskatchewan Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-2010
Record Dates: First submitted 2013-04-18; First posted 2013-04-29 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Fiber; BUN; Serum Creatinine; Uremic Symptoms; Quality of Life
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Hazard Analysis and Critical Control Points; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Foods (Placebo Comparator): For a period of 2 weeks, participants will consume control foods in addition to their usual diets.
  Interventions: Other: Control Food
- Fiber Fortified Foods (Experimental): For a period of 4 weeks, participants will consume food fortified with fiber in addition to their usual diets.
  Interventions: Other: Fiber Fortified Food

INTERVENTIONS:
Other: Control Food — For a period of 2 weeks, participants will consume control foods in addition to their usual diets.
  Other Names: Kellogg's Corn Pops; Publix Chocolate Chip Cookies; Kellogg's Special K Bar
  Arms: Control Foods
Other: Fiber Fortified Food — For a period of 4 weeks, participants will consume food fortified with fiber in addition to their usual diets.
  Other Names: Kellogg's Corn Pops with Fiber; Weight Watchers Chocolate Chip Cookies; General Mills FiberOne Bar
  Arms: Fiber Fortified Foods

SUMMARY:
A single blind, six week dietary intervention will be conducted in order to evaluate the impact of fiber fortified foods on blood urea nitrogen, kidney function and quality of life in patients presenting with a moderate to severe decline in kidney function.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) patients may consume lower than recommended amounts of dietary fiber due to typical dietary habits, dietary restrictions, and uremic symptoms. A progressive decline in kidney function causes an accumulation of uremic molecules that contribute to further progression of the disease and reduced quality of life. In an effort to evaluate the impact of added fiber on blood urea nitrogen, kidney function and quality of life in patients presenting with a moderate to severe decline in kidney function (eGFR ≤ 50 mL/min/1.73 m2), a single blind, six week dietary intervention, clinical trial will be conducted.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Be 18 years of age or older
* Have eGFR (estimated glomerular filtration rate) of less than 50 mL/min/1.73 m2 (stage 3,4 and 5 but who are not on dialysis)

Exclusion Criteria:

Participants must not:

* Have been diagnosed with acute kidney injury (AKI)
* Have been diagnosed with glumerulonephritis (GN)
* Have been on immunosuppressant/steroid medications
* Be taking a probiotic supplement and refuse to discontinue it
* Be scheduled for dialysis within 3 months of study initiation
* Have a history of liver disease
* Be on dialysis
* Have undergone renal transplantation
* Be breastfeeding
* Have active gastrointestinal bleeding
* Have a change in medications over the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Impact of added fiber on blood urea nitrogen (BUN) | up to 42 days of the study
  Blood samples (10 mL) will be taken on day 1, 14, 28, and 42. BUN will be assayed using the Urea Nitrogen Concentrated Reagent method.

SECONDARY OUTCOMES:
Impact of foods with added fiber on estimated Glomerular Filtration Rate (eGFR) | Days 1, 14, 28 and 42 of the study
  eGFR will be calculated using the Modification of Diet in Renal Disease formula on days 1, 14, 28 and 42 of the study.
Impact of foods with added fiber on Serum Creatinine | Days 1, 14, 28 and 42 of the study
  Serum creatinine will be assayed using the ADVIA Chemistry CRE_2c method.
Impact of foods with added fiber on bowel movement frequency | Daily
  Participants will complete daily diaries to evaluate bowel movement frequency.
Impact of foods with added fiber on Kidney Disease Quality of Life (KDQOL-36) questionnaire | Days 1, 14, 28 and 42
  Participants will complete the Kidney Disease Quality of Life (KDQOL-36) questionnaire for 4 specific days during the study.
Impact of foods with added fiber on Simplified Nutritional Appetite Questionnaire (SNAQ) | Days 1, 14, 28 and 42 of the study
Impact of foods with added fiber on Epworth Sleepiness Scale (ESS) | Days 1, 14, 28 and 42 of the study
Impact of foods with added fiber on Gastrointestinal Symptom Rating Scale (GSRS) | Days 1, 14, 28 and 42 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Salmean YA, Zello GA, Dahl WJ. Foods with added fiber improve stool frequency in individuals with chronic kidney disease with no impact on appetite or overall quality of life. BMC Res Notes. 2013 Dec 5;6:510. doi: 10.1186/1756-0500-6-510. PMID 24304924